CLINICAL TRIAL: NCT03878771
Title: Platelet Rich-plasma in Management of Chronic Multiple Oral Ulcers
Brief Title: PRF in Management of Chronic Multiple Oral Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Eman Magdy Ahmed, Lecturer of Oral Medicine and Dianosis, Beni-Suef University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00uad
Record Dates: First submitted 2019-03-13; First posted 2019-03-18 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Oral Ulcer Due to Pemphius Vularis; Oral Ulcer Due to Benign Mucous Membrane Pemphioid; Oral Ulcer Due to Steven Johnson's Syndrome
Keywords: Platelet rich fibrin, Oral Ulcer, Pain, Mucositis
MeSH Terms: conditions — Oral Ulcer; Pain; Mucositis | interventions — Orabase

STUDY DESIGN:
Intervention Model Description: Patients with chronic multiple oral lesions due to benign mucous membrane Pemphigoid, Pemphigus vulgaris, ans Steven Johnson's Syndrome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autologous Platelet rich fibrin in Orabase (PRF) (Experimental): applied to oral ulcer and/or mucositis 3 times per day
  Interventions: Biological: Platelet rich fibrin gel in Orabase
- Clobetasol propionate 0.05%(Dermovate cream) in orabase (Active Comparator): applied to oral ulcer and/or mucositis 3 times per day
  Interventions: Drug: Dermovate cream in Orabase

INTERVENTIONS:
Biological: Platelet rich fibrin gel in Orabase — applied on oral mucositis and /or ulcer 3 times per day
  Other Names: autologus PRF gel
  Arms: autologous Platelet rich fibrin in Orabase (PRF)
Drug: Dermovate cream in Orabase — applied on oral mucositis and /or ulcer 3 times per day
  Other Names: Clobetasol Propionate 0.05%
  Arms: Clobetasol propionate 0.05%(Dermovate cream) in orabase

SUMMARY:
PRF in orabase will be applied as a pack material on chronic oral ulcers of chronic multiple oral lesions compared to conventional topical steroid therapy with clobetasol propionate 0.05% in orabase. The outcomes measured are Pain alleviation as Primary outcome and Clinical improvement in terms of Ulcer size, Number and Mucositis score as Secondary outcomes. Time frame for outcomes assessment will be Daily for 7 Days regarding pain score and weekly for 2 weeks regarding clinical improvement.

DETAILED DESCRIPTION:
The management of oral ulcers and mucositis specially the resistant types such as oral ulcers due to auto-immune diseases is a major concern by the dentists through all the world. Topical corticosteroids, analgesics, Laser bio modulation all have been proposed as treatments with limited efficacy in many cases. There are few number of clinical trials on Plasma preparation in management of oral mucositis and oral ulcers. Platelet rich fibrin (PRF) is one of the platelet concentrates. The preparation protocol of PRF is simple and easy, could be prepared autologous and immediately placed on the oral ulcers and mucositis.

Subjects and Methods: A non Randomized clinical trial will be conducted. Ten patients with different resistant oral ulcers and mucositis were enrolled. all with grade 4 WHO mucositis score. The initial numerical ratting score of pain is 10. For all patients 20 ml blood sample will obtained in plain blood vacutainer, centrifuged for 15 minutes on 3000 rpm. The resultant gel, obtained and squeezed to prepare a membrane, the membrane will be mixed with orabase and placed over the oral ulcers and mucositis over a piece of gauze. The patients will be instructed not to eat or drink for 2 hours after application. The remaining serum after squeezing was mixed with equal amount of orabase and used topically on the oral mucositis and ulcers.

Clobetasol Propionate 0.05% in orabase will be applied to 10 control patients 3 times per day for one week.

The steps will be repeated after one week if the patients' symptomatic scores for WHO and numerical rating score were not zero.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Oral ulcers due to Benin mucous membrane pemphioid, Pemphius vulgaris and Steven Johnson's Syndrome with mucositis score 4 and pain score 10

Exclusion Criteria:

* patients with any systemic other systemic condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Pain score | 1 week
  Numerical Rating score of Pain, graded from 0 to 10, were 0 is no pain at all and 10 represent severe pain, obtaining lower values reflects improvement

SECONDARY OUTCOMES:
Mucositis | 2 weeks
  WHO mucositis score, graded from 0 to 4 were 0 no mucositis and 4 severe mucositis, obtaining lower values reflects improvement
ulcer size | 2 weeks
  Measurement in cm for the largest ulcer, expressed as maximum height x maximum width reflecting the average size, decrease in size is improvement
ulcer number | 2 weeks
  number counted for each patient, decrease in number reflects improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Eman Ahmed, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: a